CLINICAL TRIAL: NCT04491123
Title: Evaluation of Discomfort Symptoms in Patients With Refractory Cancer Pain and Intrathecal Analgesia Management
Brief Title: Intrathecal Analgesia Effects on Cancer Patients Discomfort Symptoms
Acronym: IT-ESAS
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Institut du Cancer de Montpellier - Val d'Aurelle (Other); Centre Hospitalier Universitaire de Nīmes (Other); Oncopole Toulouse (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0065
Record Dates: First submitted 2020-03-11; First posted 2020-07-29 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Refractory Cancer Pain; Intrathecal Analgesia
Keywords: Refractory cancer pain; intrathecal analgesia; pain management; discomfort symptoms management
MeSH Terms: conditions — Cancer Pain; Agnosia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Intrathecal analgesia is used in refractory cancer pain because of drug sides effects or intractable pain. The aim of this approach is to improve pain management, and also to improve patient comfort. This study will assess patient discomfort symptoms before and after setting up intrathecal analgesia.

DETAILED DESCRIPTION:
Descriptive multicenter study including patients with refractory cancer pain (unmanageable drug sides effects or intractable pain) who will receive intrathecal analgesia Patient discomfort symptoms will be evaluated before and after the beginning of intrathecal analgesia at 15, 30, 60 and 90 days.

Moreover, the impact on patient close relatives and on return home will be assessed.

ELIGIBILITY:
Inclusion criteria:

* patients aged 18 and older
* obligation of affiliation or beneficiary of a social security scheme
* patients with cancer and refractory localized cancer pain because of drug side effects or intractable pain
* localized pain in topography accessible to intrathecal analgesia (legs, abdomen and pelvis, pancoast-tobias symdrom)
* patient's informed consent for the study
* patient able to complete the evaluation questionnaires
* estimed vital prognosis more than three month
* patient with all conditions for intrathecal anagelsia

Exclusion criteria:

* patient with intracranial hypertension
* refusal of patient to be included in the study
* refusal of patient to receive intrathecal analgesia
* patient with many refractory pain localizations not accessible to intrathecal analgesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cancer patients with refractory localized cancer pain because of drug side effects or intractable pain who will receive intrathecal analgesia.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Number Evaluation of Edmonton symptoms | up to 90 days after patient inclusion
  Edmonton symptom assessment system

SECONDARY OUTCOMES:
Autonomy assessment score for activities of daily living | 1 day
  Autonomy assessment score for activities of daily living

CONTACTS AND LOCATIONS:
Overall Officials: Raphael RENAMBATZ-ICHAMBE, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC